CLINICAL TRIAL: NCT04254341
Title: Upper Airway Dilator Muscle Activity in Healthy Subjects and Patients With Obstructive Sleep Apnea During Wakefulness and Sleep
Brief Title: Dilator Muscle Activity in Health and Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, ARIE.OLIVEN, Clinical Professor, Bnai Zion Medical Center
Other Study IDs: 0096-14-BNZ
Record Dates: First submitted 2015-09-02; First posted 2020-02-05 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with OSA: Subjects that underwent regular sleep studies (PSG) and found to have moderate/severe obstructive sleep apnea
  Interventions: Other: patients with OSA
- subjects without OSA: Subjects that underwent regular PSG and found not to have sleep apnea
  Interventions: Other: patients with OSA

INTERVENTIONS:
Other: patients with OSA — Sleep study

SUMMARY:
The role of control of peri-pharyngeal muscle tone in the pathogenesis of obstructive sleep apnea (OSA) is obvious: pharyngeal obstruction occurs only during sleep; and pharyngeal collapse occurs in almost all healthy subjects during anesthesia. Better understanding of these control mechanisms may help identifying the central components of the pathogenesis of OSA.

DETAILED DESCRIPTION:
Study plan: Subjects will be studied first during wakefulness, while breathing against external resistors, to evaluate how are the peri-pharyngeal muscles recruited and activated to prevent pharyngeal collapse in the presence of negative intra-pharyngeal pressures. Thereafter, the same parameters will be evaluated during sleep, to assess muscle recruitment during intra-pharyngeal obstruction. The investigaors will record the electromyogram (EMG) of several dilator muscles, as well as the pressures above and below the area of pharyngeal collapse, and airflow.

ELIGIBILITY:
Inclusion Criteria:

1. subjects that underwent regular sleep studies and found to have either moderate/severe OSA, or no OSA.

-

Exclusion Criteria:

1. hemophilia
2. use of anti-coagulants -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult subjects with and without sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
EMG activity of peri-pharyngeal muscles during wakefulness and sleep | 4 hours
  EMG of peripharyngeal muscles will be measured during wakefulness (on external resistors) and sleep (during flow limitation), patients with OSA. EMG data will be presented as %max (0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Arie Oliven, MD, Principal Investigator — Bnai Zion

REFERENCES:
- [Background] Dotan Y, Pillar G, Schwartz AR, Oliven A. Asynchrony of lingual muscle recruitment during sleep in obstructive sleep apnea. J Appl Physiol (1985). 2015 Jun 15;118(12):1516-24. doi: 10.1152/japplphysiol.00937.2014. Epub 2015 Mar 26. PMID 25814639
- [Background] Dotan Y, Pillar G, Tov N, Oliven R, Steinfeld U, Gaitini L, Odeh M, Schwartz AR, Oliven A. Dissociation of electromyogram and mechanical response in sleep apnoea during propofol anaesthesia. Eur Respir J. 2013 Jan;41(1):74-84. doi: 10.1183/09031936.00159611. Epub 2012 May 3. PMID 22556023